CLINICAL TRIAL: NCT00000460
Title: Training Levels Comparison (TLC) Trial in Patients With Coronary Heart Disease
Brief Title: Training Levels Comparison Trial
Status: Withdrawn | Type: Observational
Why Stopped: due to lack of enrollment
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 49; R01HL037597 (NIH)
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2013-11

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Heart Diseases; Myocardial Ischemia
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Diseases; Myocardial Ischemia | interventions — High-Intensity Interval Training

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Low intensity exercise
  Interventions: Behavioral: Low intensity exercise
- High intensity exercise
  Interventions: Behavioral: High intensity exercise

INTERVENTIONS:
Behavioral: Low intensity exercise
  Groups: Low intensity exercise
Behavioral: High intensity exercise
  Groups: High intensity exercise

SUMMARY:
To determine the effects of high or low intensity long-term exercise conditioning in patients with coronary artery disease.

DETAILED DESCRIPTION:
BACKGROUND:

A vast amount of literature exists on the improvements in work capacity, reduction of risk factors, and an increased feeling of well-being among coronary heart disease patients after physical training programs. Previous observations of short-term training programs which resulted in an increase in physical working capacity have not usually shown a cardiac change. The National Exercise and Heart Disease Project did not show such changes, but the exercise level may have been inadequate. Several other studies suggested that more prolonged and intense training could result in improved cardiac function.

DESIGN NARRATIVE:

Patients were randomized to high intensity or low intensity long-term exercise groups. Compliance was strengthened by randomizing following a sequence of eligibility visits and after a test period of subject reaction to an exercise program. The primary endpoint was change in exercise ejection fraction at one year. Secondary endpoints included changes in lipid levels, body composition, blood pressure and heart rate measurements, glucose tolerance, quality of life measures, compliance, and progression of disease. Patients were classified into one of four strata based on the documented history of myocardial infarction and resting left ventricular ejection fraction. Within each stratum, patients were assigned in equal numbers to the two intensity levels of exercise intervention. All exercise prescriptions were based on exercise testing of patients maintained on their usual medical regimen including drugs. Patients underwent standardized multistage treadmill exercise testing monitored by Doppler echocardiogram at baseline, just prior to randomization and at the three month, six month, one year and two year visits. Patients participated in the structured group exercise sessions three days per week. Each exercise session was preceded by and ended with a five to fifteen minute warm-up and cool-down session. Each patient was given an exercise prescription that included a 30 minute period of walking or of walking and jogging sequences and 15 minutes of arm-leg bicycle ergometer exercise. Recruitment started in May 1987. The last patient was enrolled in March 1990.

ELIGIBILITY:
Men, ages 30 to 67, with documented coronary heart disease.

Ages: 30 Years to 67 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men between the ages of 30 and 67 who respond to an advertisement for research participants.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 1986-12; Primary Completion 1991-03 (Actual); Study Completion 1991-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Albert Oberman, Principal Investigator — University of Alabama at Birmingham

REFERENCES:
- [Background] Lee JY, Oberman A, Fletcher GF, Raczynski JM, Fletcher BJ, Nanda NC, Jensen BE. Design of the training levels comparison trial. Control Clin Trials. 1994 Feb;15(1):59-76. doi: 10.1016/0197-2456(94)90028-0. PMID 8149771
- [Background] Kim JR, Oberman A, Fletcher GF, Lee JY. Effect of exercise intensity and frequency on lipid levels in men with coronary heart disease: Training Level Comparison Trial. Am J Cardiol. 2001 Apr 15;87(8):942-6; A3. doi: 10.1016/s0002-9149(01)01425-4. PMID 11305982
- [Background] Jensen BE, Fletcher BJ, Rupp JC, Fletcher GF, Lee JY, Oberman A. Training level comparison study. Effect of high and low intensity exercise on ventilatory threshold in men with coronary artery disease. J Cardiopulm Rehabil. 1996 Jul-Aug;16(4):227-32. doi: 10.1097/00008483-199607000-00003. PMID 8872288
- [Background] Lee JY, Jensen BE, Oberman A, Fletcher GF, Fletcher BJ, Raczynski JM. Adherence in the training levels comparison trial. Med Sci Sports Exerc. 1996 Jan;28(1):47-52. doi: 10.1097/00005768-199601000-00013. PMID 8775354